CLINICAL TRIAL: NCT04072432
Title: A Phase 1b Dose-escalating Study With RBT-3 in Healthy Volunteers and Volunteers With Chronic Kidney Disease Stage 3/4
Brief Title: A Study of RBT-3 in Healthy Volunteers and Volunteers With Stage 3/4 Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REN-002
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2020-03-03 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 120 mg (Experimental)
  Interventions: Drug: RBT-3
- 240 mg (Experimental)
  Interventions: Drug: RBT-3
- 360 mg (Experimental)
  Interventions: Drug: RBT-3

INTERVENTIONS:
Drug: RBT-3 — intravenous administration

SUMMARY:
This is a Phase 1b, single center, dose-escalating study evaluating the safety, tolerability, and pharmacodynamic effect of RBT-3 in healthy volunteers and in subjects with stage 3-4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 to 80 years (inclusive, at time of ICF).
2. Body weight <125 kg.
3. Able and willing to comply with all study procedures.
4. Female subjects must be either post-menopausal for at least 1 year or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from Screening until 8 days after study drug administration.

   Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from screening until 8 days after study drug administration. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.
5. CKD as determined by estimated glomerular filtration rate (eGFR) between 15-59 ml/min as estimated using the CKD-EPI equation (CKD class 3-4).

Exclusion Criteria:

1. History of malignancy except carcinoma in situ in the cervix, early stage prostate cancer or non-melanoma skin cancers.
2. Use of investigational drugs or participation in another clinical trial within 30 days or 5 half-lives prior to screening, whichever is longer.
3. Serum ferritin > 500 ng/ml or who have received IV iron within 28 days of screening.
4. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
5. Any significant acute or chronic diseases, excluding CKD (eGFR ≥15 ml/min).
6. Regular use of drugs of abuse and/or positive findings on urinary drug screening.
7. Current tobacco use and/or positive findings on urinary cotinine screening.
8. Subjects who are severely physically or mentally incapacitated and who, in the opinion of investigator, are unable to perform the subjects' tasks associated with the protocol.
9. Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
10. Known hypersensitivity or previous anaphylaxis to FeS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside Clinical Research, Edgewater, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 120 mg; 240 mg; 360 mg: Single IV infusion
Period: Overall Study
Arm/Group | 120 mg | 240 mg | 360 mg
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 120 mg | 240 mg | 360 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (7.32) | 57.7 (14.87) | 63.3 (11.83) | 60.3 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 10
  Male | 2 | 2 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 5 | 4 | 3 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Effect of RBT-3 on Plasma Ferritin Levels
Time Frame: 24 hours post-infusion
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio (24 h post-infusion over baseline)
Arm/Group | 120 mg | 240 mg | 360 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio (24 h post-infusion over baseline) | 2.49 [1.94 to 3.19] | 4.42 [3.45 to 5.66] | 4.90 [3.82 to 6.28]

2. Primary Outcome: Effect of RBT-3 on Plasma HO-1 Levels
Time Frame: 24 hours post-infusion
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio (24 h post-infusion over baseline)
Arm/Group | 120 mg | 240 mg | 360 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio (24 h post-infusion over baseline) | 0.0171 [-0.694 to 0.728] | -0.7086 [-1.419 to 0.002] | -0.0641 [-0.775 to 0.646]

ADVERSE EVENTS:
Time Frame: 8 days
Arm/Group | 120 mg | 240 mg | 360 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 120 mg (N=6) | 240 mg (N=6) | 360 mg (N=6)
Mild Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04072432/Prot_004.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT04072432/SAP_005.pdf